CLINICAL TRIAL: NCT06580210
Title: Prospective Multicenter Clinical Investigation to Evaluate the Performance and the Safety of the Mechanical Decongestant Seawater Spray Enriched With Essential Oils From Laboratoires Gilbert (DEMECA)
Brief Title: Performance and Safety Assessment of the Mechanical Decongestant Seawater Spray Enriched With Essential Oils From Laboratoires Gilbert in Patient With Acute Rhinitis Associated With Nasal Obstruction
Acronym: DEMECA
Status: Recruiting | Type: Observational
Sponsor: Laboratoires Gilbert (Industry)
Collaborators: EVAMED (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A01585-38
Record Dates: First submitted 2024-08-29; First posted 2024-08-30 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Acute Rhinitis; Nasal Obstruction; Rhinosinusitis; Rhinopharyngitis; Allergic Rhinitis
MeSH Terms: conditions — Common Cold; Nasal Obstruction; Rhinosinusitis; Nasopharyngitis; Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this post-market clinical investigation is to assess the performance and the safety of the mechanical decongestant seawater spray enriched with essential oils from Laboratoires Gilbert. The study will evaluate the results of the spray on the acute rhinitis with nasal obstruction over a 7 days period.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient ≥ 12 years,
* 2. Patient with acute rhinitis associated with nasal obstruction during infectious episodes such as rhynopharyngitis (cold), rhinosinusitis, or during non-infectious episodes as allergic rhinitis,
* 3. a. Informed adult patient who has given written consent prior to any study specific procedure,
* b. Informed minor patients who has given assent and whose legal guardians have given written consent prior to any study specific procedure,
* 4. Patient able to meet the study requirements (questionnaire completion),
* 5. Patient affiliated to a social security scheme.

Exclusion Criteria:

* 1. Patient who does not want to participate to the clinical investigation,
* 2. Hypersensitivity to seawater and/or known allergies to any of the ingredients of the spray,
* 3. A child with a history of febrile convulsions,
* 4. Diseases leading to respiratory insufficiency,
* 5. Patient suffering from nasal deformity or nasal polyps leading to chronic nasal obstruction,
* 6. Patient on local ans systemic vasoconstrictors, local and systemic corticosteroids and antihistamines, non-steroidal anti-inflammatory (NSAIDs), antibiotics and local antiseptics,
* 7. Concomitant use of other nasal sprays, essential oils for local nasal use and nsal cream or gel,
* 8. Patient under guardianship, curatorship of safeguard of justice.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participation in the study is open to patients who buy the mechanical decongestant seawater spray on request or on the advice of their pharmacist. Patients are offered the opportunity to take part in the clinical investigation at the time of payment and after the eligibility critera have been checked by the pharmacist.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-07 (Estimated)

PRIMARY OUTCOMES:
Performance of the mechanical decongestant seawater spray enriched with essential oils from Laboratoires Gilbert at 3 days | From Day 0 to Day 3
  Proportion of patients presenting a change of the symptom -nasal obstruction- by at least 1 pt, in the SNOT22 Test (item 22), between Day 0 (at inclusion in the pharmacy before using the spray) and Day 3 (in the evening after the last daily use of the spray). This item is scaled form 0 to 5 and 5 is the worst value.

SECONDARY OUTCOMES:
Performance of the mechanical decongestant seawater spray enriched with essential oils from Laboratoires Gilbert after the first use | At Day 0
  Proportion of patients who experienced an amelioration of their nasal obstruction after the first use of the spray at Day 0 on patient questionnaire.
Subjective feeling of reduced nasal obstruction on each day of use | From Day 0 and Day 6
  Proportion of patients with a reduction in the symptom -nasal obstruction- of at least 1pt, in the SNOT22 Test (item 22), on each day of use (between Day 0 and Day 6). The item is scaled form 0 to 5 and 5 is the worst value.
Subjective feeling of nasal secretion thinning on each day of use | From Day 0 to Day 6
  Proportion of patients presenting a change of the symptom -thick nasal discharge- by at least 1 pt, in the SNOT22 Test, and on each day of use (from Day 0 to Day 6)
Subjective feeling of nasal cavity cleansing (freshness) on each day of use | From Day 0 to Day 6
  Proportion of patients who experienced nasal cavity cleansing (feeling of freshness), on Patient Questionnaire, and on each day of use (from Day 0 to Day 6).
Subjective feeling of relief of nasal irritation (mucous membrane) on each day of use | From Day 0 to Day 6
  Proportion of patients who experienced relief of nasal irritation (mucous membrane), on Patient Questionnaire, on each day of use (from Day 0 to Day 6).
Subjective feeling of relief of nasal itching on each day of use | From Day 0 to Day 6
  Proportion of patients who experienced relief of nasal itching, on Patient Questionnaire, on each day of use (from Day 0 to Day 6).
Subjective feeling of nasal cavity cleansing (freshness) immediately (2 minuts) after the use of the spray at Day 0 | At Day 0 and Day 6
  Proportion of patient who experienced nasal cavity cleansing (feeling of freshness) immediately (2 minuts) after the use of the spray, on Patient Questionnaire, at Day 0 and Day 6.
Subjective feeling of reduced nasal obstruction immediately (2 minuts) after the use of the spray at Day 6 | At Day 6
  Proportion of patient who experienced a reduction of nasal obstruction immediately (2 minuts) after the use of the spray, on Patient Questionnaire, at Day 6.
Subjective feeling of reduced nasal obstruction immediately (2 minuts) after the use of the spray at Day 0 | At Day 0
  Proportion of patient who experienced a reduction of nasal obstruction immediately (2 minuts) after the use of the spray, on Patient Questionnaire, at Day 0.
Improvement in the patient s quality of life after 7 days of use | At Day 0 et Day 6
  Proportion of patients who experienced an improvement in quality of life, on Patient Questionnaire (scale of 0-10 with 10 is the best value), between Day 0 and Day 6.
Patient satisfaction with the spray after 7 days of use | At Day 6
  Proportion of patients satisfied with the spray on a 4-points scale, at Day 6. The best value is -very satisfied- and the worst value is -very unsatisfied-.
Patient s recommendation of the spray after 7 days of use | At Day 6
  Proportion of patients who would recommend the spray, on a 4-points scale, at Day 6. The best value is -definitely yes- and the worst value is -definitely no-.
Patient s willingness to continue using the spray at Day 6 | At day 6
  Proportion of patients who will continue to use the spray and the reason if he does not want to continue, on a 4-points scale, at Day 6. The best value is -definitely yes- and the worst value is -definitely no-.
Facility of use of the spray after 7 days of use | At Day 6
  Proportion of patients who find the spray easy to use, on a 4-points scale, at Day 6. The best value is -very easy- and the worst value is -very difficult-.
Evolution of the overall severity of symptoms | At Day 0 and Day 3
  Average SNOT22 score each day and comparison of SNOT22 score at Day 3 versus DAy 0 (baseline). [0 to 220] with 0 is the best value and 220 is the worst value.
Sensations of tingling and transient irritation | From Day 0 to Day 6
  Proportion of patients with at least 1 adverse event among :
  * tingling sensation
  * sensations of transient irritation during the 7 days of use.
All device deficiencies reported by patients using the spray during the 7 days of use | From Day 0 to Day 6
  Proportion of patients with at least 1 device deficiency during the clinical investigation.
All adverse events reported by patients using the spray during the 7 days of use | From Day 0 to Day 6
  All adverse events reported by the patient during the clinical investigation.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Pharmacie du Pont Saint Jean, Bayeux
  - Pharmacie de la Guérinière, Caen
  - Pharmacie de la Force, La Force

IPD SHARING:
Plan to Share IPD: No